CLINICAL TRIAL: NCT00860119
Title: Open-Label, Randomized, Single-Dose, 2-Way Crossover Pivotal Bioequivalence Study Comparing Alprazolam Immediate Release (IR) Tablets (Administered Orally) And Alprazolam Sublingual (SL) Tablets (Administered Sublingually)
Brief Title: Bioequivalence of Alprazolam Sublingual vs Oral Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131017
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Bioequivalence, Pharmacokinetics, Alprazolam, Sublingual
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sublingual tablet (Experimental): Test treatment
  Interventions: Drug: alprazolam sublingual tablet
- Oral tablet (Experimental): Reference treatment
  Interventions: Drug: alprazolam oral tablet

INTERVENTIONS:
Drug: alprazolam sublingual tablet — 1 mg alprazolam sublingual tablet, given as a single dose to each subject
  Arms: Sublingual tablet
Drug: alprazolam oral tablet — 1 mg alprazolam immediate release oral tablet, given as a single dose to each subject
  Other Names: Xanax
  Arms: Oral tablet

SUMMARY:
This study tests the assumption that the bioavailability of alprazolam from a new sublingual formulation is the same as that from a standard orally administered tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* BMI 17.5 - 30.5
* Must provide informed consent

Exclusion Criteria:

* Clinically significant disease
* Narrow angle glaucoma
* Positive drug screen

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Alprazolam bioavailability assessed as area under the concentration-time curve (AUC) and maximum concentration (Cmax) | 11 days

SECONDARY OUTCOMES:
Alprazolam time of maximum concentration (Tmax) and half life | 11 days
Adverse events, clinical laboratory tests, vital signs | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ahmedabad, Gujarat, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131017&StudyName=Bioequivalence%20of%20alprazolam%20sublingual%20vs%20oral%20tablets